CLINICAL TRIAL: NCT02700984
Title: An Observational Multicenter Clinical Study to Assess the Long-Term Safety of the CyPass Micro-Stent in Patients With Primary Open Angle Glaucoma Who Have Completed Participation in the COMPASS Trial
Brief Title: A Study to Assess Long-Term Safety of the CyPass Micro-Stent in Patients Completing the COMPASS Trial
Acronym: COMPASS-XT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Transcend Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TMI-09-01-E; GLD122b-C001 (Other: Alcon)
Record Dates: First submitted 2016-02-28; First posted 2016-03-07 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2019-05

CONDITIONS: Primary Open Angle Glaucoma (POAG)
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cataract Surgery + CyPass (Experimental): CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial)
  Interventions: Device: CyPass Micro-Stent; Procedure: Cataract Surgery
- Cataract Surgery Only (Active Comparator): Cataract Surgery (COMPASS trial) with no CyPass Micro-Stent implantation
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Device: CyPass Micro-Stent — The CyPass Micro-Stent is a small tube with a through-lumen designed to redirect aqueous fluid from the front into the back of the eye. The device is implanted after completion of cataract surgery.
  Arms: Cataract Surgery + CyPass
Procedure: Cataract Surgery — Cataract surgery involves the removal of the natural lens, which has become clouded (called a cataract), and insertion of an artificial lens (called an intraocular lens). This procedure is done through a small surgical incision in the eye.

SUMMARY:
The purpose of this study is to evaluate the long-term safety of the CyPass Micro-Stent in subjects who completed Study Protocol TMI-09-01, COMPASS Trial.

DETAILED DESCRIPTION:
The COMPASS Trial (TMI-09-01) was a prospective, randomized, comparative multicenter study to assess the safety and effectiveness of the CyPass Micro-Stent in subjects with primary open angle glaucoma who were undergoing cataract surgery. In the study, 505 subjects were randomized to either the CyPass group, who underwent cataract surgery and received the CyPass Micro-Stent, or the Control group, who underwent cataract surgery alone. All subjects randomized were to be followed for 2 years postoperatively. Four hundred eighty (480) subjects completed this study.

The COMPASS-XT (TMI-09-01-E) Trial is designed to collect safety data beyond 24 months postoperatively for subjects who completed the COMPASS Trial. In COMPASS-XT, clinical data will be collected at 36 months, 48 months, and 60 months postoperatively for a total of 5 year follow-up across the 2 studies.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the COMPASS Trial
2. Understands study requirements and is willing to follow study instructions and return for study visits

Exclusion Criteria:

1. Systemic disease that would put subject health at risk and/or prevent completion of required study visits.
2. Early termination from the COMPASS Trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, Research, Study Director — Alcon Research
Locations (22):
- United States (22):
  - Alcon Investigative Site, Glendale, Arizona
  - Alcon Investigative Site, Fayetteville, Arkansas
  - Alcon Investigative Site, La Jolla, California
  - Alcon Investigative Site, Orange, California
  - Alcon Investigative Site, Fort Collins, Colorado
  - Alcon Investigative Site, Parker, Colorado
  - Alcon Investigative Site, Boynton Beach, Florida
  - Alcon Investigative Site, Cape Coral, Florida
  - Alcon Investigative Site, Sioux City, Iowa
  - Alcon Investigative Site, Garden City, Kansas
  - Alcon Investigative Site, Boston, Massachusetts
  - Alcon Investigative Site, St Louis, Missouri
  - Alcon Investigative Site, Vineland, New Jersey
  - Alcon Investigative Site, Cincinnati, Ohio
  - Alcon Investigative Site, Oklahoma City, Oklahoma
  - Alcon Investigative Site, Kingston, Pennsylvania
  - Alcon Investigative Site, West Mifflin, Pennsylvania
  - Alcon Investigative Site, Maryville, Tennessee
  - Alcon Investigative Site, Nashville, Tennessee
  - Alcon Investigative Site, Dallas, Texas
  - Alcon Investigative Site, Fort Worth, Texas
  - Alcon Investigative Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 23 study sites located in the US.
Pre-assignment Details: This reporting group includes all enrolled subjects (282).
Period: Overall Study
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Started (All enrolled subjects) | 215 | 67
Completed (All subjects who completed the 60-month assessment) | 200 | 53
Not Completed | 15 | 14
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Reason not specified | 3 | 2

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only | Total
Number analyzed (Participants) | 215 | 67 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (7.9) | 70.8 (7.5) | 69.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 37 | 153
  Male | 99 | 30 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 204 | 63 | 267
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 191 | 58 | 249
  Black or African American | 21 | 7 | 28
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Missing | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 5-year Annualized Rate (Percentage) of Sight-threatening Adverse Events, by Treatment Group
Description: Sight-threatening adverse events occurring in the study eye included, but were not limited to: BCVA loss of ≥ 3 lines, endophthalmitis, corneal decompensation, severe retinal detachment, severe choroidal hemorrhage, severe choroidal detachment and aqueous misdirection. The number of events at the end of Year 5 was divided by the number of eyes at risk at the beginning of Year 1 for a 5-year annualized rate. The 5-year annualized rate is reported as a percentage, with the last annual non-censored rate divided by 5. Inferential testing was not planned for this endpoint.
Time Frame: Up to Month 60 postoperative
Population: All enrolled subjects with available data
Measure: Number (95% Confidence Interval); unit: rate (percentage) of adverse events
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
Number analyzed (eyes) | 215 | 67
rate (percentage) of adverse events | 0.19 [0.05 to 0.76] | 0.30 [0.04 to 2.03]

2. Secondary Outcome: Number of Subjects According to Best Corrected Visual Acuity (BCVA) by Visit
Description: Best corrected (with spectacles or other visual corrective devices) VA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) charts at 1 or 4 meters and determined by total number of letters read correctly. 20/20 Snellen is considered 'normal' vision. A larger denominator indicates a lower visual acuity. Baseline, Month 12, and Month 24 data derived from previous COMPASS trial. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Baseline, Month 12, 24, 36, 48, 60 postoperative
Population: All enrolled subjects with available data
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
subjects
  20/20 or Better @ Baseline | 14 | 2
  20/25 or Better @ Baseline | 55 | 17
  20/32 or Better @ Baseline | 106 | 34
  20/40 or Better @ Baseline | 171 | 52
  Worse than 20/40 @ Baseline | 44 | 15
  20/20 or Better @ Month 12: number analyzed (Participants) | 214 | 66
  20/20 or Better @ Month 12 | 145 | 49
  20/25 or Better @ Month 12: number analyzed (Participants) | 214 | 66
  20/25 or Better @ Month 12 | 192 | 59
  20/32 or Better @ Month 12: number analyzed (Participants) | 214 | 66
  20/32 or Better @ Month 12 | 212 | 64
  20/40 or Better @ Month 12: number analyzed (Participants) | 214 | 66
  20/40 or Better @ Month 12 | 213 | 66
  Worse than 20/40 @ Month 12: number analyzed (Participants) | 214 | 66
  Worse than 20/40 @ Month 12 | 1 | 0
  20/20 or Better @ Month 24 | 150 | 46
  20/25 or Better @ Month 24 | 198 | 60
  20/32 or Better @ Month 24 | 213 | 63
  20/40 or Better @ Month 24 | 215 | 66
  Worse than 20/40 @ Month 24 | 0 | 1
  20/20 or Better @ Month 36: number analyzed (Participants) | 134 | 43
  20/20 or Better @ Month 36 | 72 | 27
  20/25 or Better @ Month 36: number analyzed (Participants) | 134 | 43
  20/25 or Better @ Month 36 | 105 | 34
  20/32 or Better @ Month 36: number analyzed (Participants) | 134 | 43
  20/32 or Better @ Month 36 | 121 | 42
  20/40 or Better @ Month 36: number analyzed (Participants) | 134 | 43
  20/40 or Better @ Month 36 | 132 | 43
  Worse than 20/40 @ Month 36: number analyzed (Participants) | 134 | 43
  Worse than 20/40 @ Month 36 | 2 | 0
  20/20 or Better @ Month 48: number analyzed (Participants) | 174 | 52
  20/20 or Better @ Month 48 | 102 | 33
  20/25 or Better @ Month 48: number analyzed (Participants) | 174 | 52
  20/25 or Better @ Month 48 | 143 | 43
  20/32 or Better @ Month 48: number analyzed (Participants) | 174 | 52
  20/32 or Better @ Month 48 | 165 | 50
  20/40 or Better @ Month 48: number analyzed (Participants) | 174 | 52
  20/40 or Better @ Month 48 | 172 | 52
  Worse than 20/40 @ Month 48: number analyzed (Participants) | 174 | 52
  Worse than 20/40 @ Month 48 | 2 | 0
  20/20 or Better @ Month 60: number analyzed (Participants) | 196 | 51
  20/20 or Better @ Month 60 | 126 | 33
  20/25 or Better @ Month 60: number analyzed (Participants) | 196 | 51
  20/25 or Better @ Month 60 | 165 | 45
  20/32 or Better @ Month 60: number analyzed (Participants) | 196 | 51
  20/32 or Better @ Month 60 | 185 | 50
  20/40 or Better @ Month 60: number analyzed (Participants) | 196 | 51
  20/40 or Better @ Month 60 | 192 | 51
  Worse than 20/40 @ Month 60: number analyzed (Participants) | 196 | 51
  Worse than 20/40 @ Month 60 | 4 | 0

3. Secondary Outcome: Number of Subjects Who Reported at Least One Protocol-specified Ocular Adverse Event in the Study Eye
Description: Ocular adverse events in the study eye could include, but were not limited to, BCVA loss of 2 lines (10 letters) or more on the ETDRS chart in comparison with the best BCVA reported in Study Protocol TMI-09-01, endophthalmitis, corneal edema, and corneal decompensation. Inferential testing was not planned for this endpoint.
Time Frame: Up to Month 60 postoperative
Population: All enrolled subjects
Measure: Number; unit: Subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
Subjects | 60 | 13

4. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Corneal Edema
Description: Corneal Edema (swelling of the cornea) was assessed by the investigator during slit-lamp examination and rated on a 4-point scale: None (transparent and clear or less than mild), Mild (dull glassy appearance), Moderate (Dull glassy appearance of epithelium with large number of vacuoles), and Severe (epithelial bullae and/or stromal edema, localized or diffuse, with or without stromal striae). Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 168 | 50
  None at Month 36 | 167 | 50
  Mild at Month 36: number analyzed (Participants) | 168 | 50
  Mild at Month 36 | 1 | 0
  None at Month 48: number analyzed (Participants) | 190 | 55
  None at Month 48 | 190 | 55
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 199 | 53
  Mild at Month 60: number analyzed (Participants) | 200 | 53
  Mild at Month 60 | 1 | 0

5. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Corneal Staining/Erosion
Description: Corneal Staining (appearance of tissue disruption and other pathophysiological changes) and erosion (abrasion) were assessed by the investigator during slit-lamp examination and rated on a 4-point scale: None (no fluorescein staining of epithelium, OR less than mild), Mild (slight fluorescein staining confined to a small focus), Moderate (regionally dense fluorescein staining (1 mm or greater in diameter) with underlying structure moderately visible), and Severe (marked fluorescein staining or epithelial loss). Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 168 | 50
  None at Month 36 | 159 | 48
  Mild at Month 36: number analyzed (Participants) | 168 | 50
  Mild at Month 36 | 8 | 2
  Moderate at Month 36: number analyzed (Participants) | 168 | 50
  Moderate at Month 36 | 1 | 0
  None at Month 48: number analyzed (Participants) | 190 | 55
  None at Month 48 | 181 | 52
  Mild at Month 48: number analyzed (Participants) | 190 | 55
  Mild at Month 48 | 8 | 3
  Moderate at Month 48: number analyzed (Participants) | 190 | 55
  Moderate at Month 48 | 1 | 0
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 191 | 51
  Mild at Month 60: number analyzed (Participants) | 200 | 53
  Mild at Month 60 | 6 | 2
  Moderate at Month 60: number analyzed (Participants) | 200 | 53
  Moderate at Month 60 | 3 | 0

6. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Anterior Chamber Cells
Description: Inflammatory anterior chamber cells (cells in the front portion of the eye) were assessed by the investigator during slit-lamp examination and reported in one of 6 categories according to cells per 1x1 mm slit: 0-<1 cell, 1-5 cells, 6-15 cells, 16-25 cells, and 26-50 cells, and >50 cells. Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  0 - < 1 cell at Month 36: number analyzed (Participants) | 168 | 50
  0 - < 1 cell at Month 36 | 168 | 50
  0 - < 1 cell at Month 48: number analyzed (Participants) | 190 | 55
  0 - < 1 cell at Month 48 | 189 | 55
  1 - 5 cells at Month 48: number analyzed (Participants) | 190 | 55
  1 - 5 cells at Month 48 | 1 | 0
  0 - < 1 cell at Month 60: number analyzed (Participants) | 200 | 53
  0 - < 1 cell at Month 60 | 200 | 53

7. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Anterior Chamber Flare
Description: Anterior Chamber Flare (protein escaping from dilated vessels) was assessed by the investigator during slit-lamp examination and rated on a 5-point scale: None, Faint, Moderate (iris and lens details clear), Marked (iris and lens details hazy), and Intense (fibrin or plastic aqueous). The presence of flare is a sign of intraocular inflammation. Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 168 | 50
  None at Month 36 | 168 | 50
  None at Month 48: number analyzed (Participants) | 190 | 55
  None at Month 48 | 190 | 55
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 200 | 53

8. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Iris Atrophy/Erosion
Description: Iris Atrophy/Erosion (deterioration) was assessed by the investigator during slit-lamp examination and rated on a 4-point scale: None, Mild, Moderate, and Severe. Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 164 | 50
  None at Month 36 | 163 | 49
  Mild at Month 36: number analyzed (Participants) | 164 | 50
  Mild at Month 36 | 1 | 1
  None at Month 48: number analyzed (Participants) | 190 | 55
  None at Month 48 | 189 | 55
  Mild at Month 48: number analyzed (Participants) | 190 | 55
  Mild at Month 48 | 1 | 0
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 198 | 53
  Mild at Month 60: number analyzed (Participants) | 200 | 53
  Mild at Month 60 | 2 | 0

9. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Iris Peaking
Description: Iris Peaking (one part of the iris pulled to a peak resulting in an irregular pupil) was assessed by the investigator during slit-lamp examination and rated on a 4-point scale: None, Mild, Moderate, and Severe. Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 164 | 50
  None at Month 36 | 163 | 50
  Mild at Month 36: number analyzed (Participants) | 164 | 50
  Mild at Month 36 | 1 | 0
  None at Month 48: number analyzed (Participants) | 189 | 55
  None at Month 48 | 188 | 55
  Mild at Month 48: number analyzed (Participants) | 189 | 55
  Mild at Month 48 | 1 | 0
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 200 | 53

10. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Iris Rubeosis
Description: Iris Rubeosis (abnormal blood vessels (formed by neovascularization) found on the surface of the iris) was assessed by the investigator during slit-lamp examination and rated on a 4-point scale: None, Mild, Moderate, and Severe. Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 164 | 50
  None at Month 36 | 164 | 50
  None at Month 48: number analyzed (Participants) | 190 | 55
  None at Month 48 | 190 | 55
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 200 | 53

11. Secondary Outcome: Slit-lamp Examination Results at Visits 36, 48, and 60, by Treatment Group - Posterior Capsule Opacification (PCO) Severity
Description: PCO (cloudy layer of scar tissue behind the lens implant) Severity was assessed by the investigator during slit-lamp examination and rated on a 6-point scale: None, Minimal, Mild, Moderate, Severe, and Unspecified. Only the categories with reported data are included. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: All subjects with available data at that visit
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 200 | 55
subjects
  None at Month 36: number analyzed (Participants) | 166 | 49
  None at Month 36 | 114 | 42
  Minimal at Month 36: number analyzed (Participants) | 166 | 49
  Minimal at Month 36 | 27 | 3
  Mild at Month 36: number analyzed (Participants) | 166 | 49
  Mild at Month 36 | 17 | 2
  Moderate at Month 36: number analyzed (Participants) | 166 | 49
  Moderate at Month 36 | 5 | 2
  Unspecified at Month 36: number analyzed (Participants) | 166 | 49
  Unspecified at Month 36 | 3 | 0
  None at Month 48: number analyzed (Participants) | 190 | 55
  None at Month 48 | 132 | 43
  Minimal at Month 48: number analyzed (Participants) | 190 | 55
  Minimal at Month 48 | 29 | 8
  Mild at Month 48: number analyzed (Participants) | 190 | 55
  Mild at Month 48 | 25 | 4
  Moderate at Month 48: number analyzed (Participants) | 190 | 55
  Moderate at Month 48 | 4 | 0
  None at Month 60: number analyzed (Participants) | 200 | 53
  None at Month 60 | 138 | 41
  Minimal at Month 60: number analyzed (Participants) | 200 | 53
  Minimal at Month 60 | 32 | 7
  Mild at Month 60: number analyzed (Participants) | 200 | 53
  Mild at Month 60 | 26 | 4
  Moderate at Month 60: number analyzed (Participants) | 200 | 53
  Moderate at Month 60 | 4 | 1

12. Secondary Outcome: Gonioscopy at Visits 36, 48, and 60, CyPass Subjects Only
Description: For subjects in the CyPass group, gonioscopic examination was performed to assess the position of the CyPass Micro-Stent in the angle and with respect to the iris and the corneal endothelium. A visible CyPass Micro-Stent indicated a lack of adhesions (favorable). One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: Number of eyes with available data and CyPass not explanted before visit
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- CyPass Visible: CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial) and visible by gonioscopy
- Cypass Not Visible: CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial) and not visible by gonioscopy
Arm/Group | CyPass Visible | Cypass Not Visible
Number analyzed (Participants) | 177 | 177
Number analyzed (eyes) | 177 | 177
eyes
  Month 36: number analyzed (eyes) | 48 | 48
  Month 36 | 47 | 1
  Month 48: number analyzed (eyes) | 140 | 140
  Month 48 | 133 | 7
  Month 60 | 162 | 15

13. Secondary Outcome: Number of Subjects With Clinically Significant Findings Noted During Fundus Examinations
Description: The dilated fundus examination was performed by the investigator to evaluate the health of the vitreous, retina, macula, choroid, and optic nerve. Clinically significant findings are reported categorically. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 36, 48, 60 postoperative
Population: Subjects with available data at each visit
Measure: Number; unit: subjects
Groups:
- Cataract Surgery + CyPass, Month 36; Cataract Surgery + CyPass, Month 48; Cataract Surgery + CyPass, Month 60: CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial)
- Cataract Surgery Only, Month 36; Cataract Surgery Only, Month 48; Cataract Surgery Only, Month 60: Cataract surgery (COMPASS trial) with no CyPass Micro-Stent implantation
Arm/Group | Cataract Surgery + CyPass, Month 36 | Cataract Surgery + CyPass, Month 48 | Cataract Surgery + CyPass, Month 60 | Cataract Surgery Only, Month 36 | Cataract Surgery Only, Month 48 | Cataract Surgery Only, Month 60
Number analyzed (Participants) | 103 | 168 | 196 | 26 | 44 | 49
subjects
  Dry age-related macular degeneration: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Dry age-related macular degeneration | 0 | 0 | 1 |  |  |
  Glaucomatous optic disc atrophy | 1 | 3 | 2 | 0 | 1 | 1
  Macular degeneration: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Macular degeneration | 0 | 0 | 1 |  |  |
  Macular fibrosis: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Macular fibrosis | 0 | 1 | 1 |  |  |
  Macular hole: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Macular hole | 0 | 0 | 1 |  |  |
  Macular oedema: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Macular oedema | 0 | 1 | 1 |  |  |
  Neovascular age-related macular degeneration: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Neovascular age-related macular degeneration | 0 | 1 | 0 |  |  |
  Optic atrophy: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Optic atrophy | 0 | 0 | 1 |  |  |
  Optic nerve disorder: number analyzed (Participants) | 103 | 168 | 196 | 0 | 0 | 0
  Optic nerve disorder | 2 | 1 | 1 |  |  |
  Retinal drusen | 0 | 0 | 1 | 1 | 1 | 0
  Retinal haemorrhage: number analyzed (Participants) | 0 | 0 | 0 | 26 | 44 | 49
  Retinal haemorrhage |  |  |  | 0 | 1 | 0

14. Secondary Outcome: Change From Month 24 in Visual Field Mean Deviation
Description: Visual field (how much one can see to each side while focusing the eyes on a central point (peripheral vision)) deviations were obtained with a Humphrey automated perimeter using the 24-2 SITA standard testing method. Normal deviation values are typically within 0 to -2 decibels (dB) and become more negative as the overall field worsens. Month 24 data derived from COMPASS trial. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 24, 36, 48, 60 postoperative
Population: All subject eyes for which data was available at the visit
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 66
dB
  Month 24 | -2.8 (3.3) | -3.2 (4.0)
  Change at Month 36: number analyzed (Participants) | 58 | 17
  Change at Month 36 | -0.0 (2.6) | -0.2 (1.5)
  Change at Month 48: number analyzed (Participants) | 142 | 41
  Change at Month 48 | -0.7 (2.3) | -0.2 (2.3)
  Change at Month 60: number analyzed (Participants) | 181 | 47
  Change at Month 60 | -0.8 (3.6) | -0.6 (2.2)

15. Secondary Outcome: Change From Month 24 in Central Corneal Thickness
Description: Central corneal thickness was evaluated by Pachymetry and measured in micrometers (μm). A negative number indicates a decrease in corneal thickness (unfavorable). Month 24 data derived from COMPASS trial. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Month 24, 36, 48, 60 postoperative
Population: Subject eyes for which data was available at the visit
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
micrometers
  Month 24 | 553.8 (35.1) | 558.1 (31.9)
  Change at Month 36: number analyzed (Participants) | 23 | 8
  Change at Month 36 | 4.7 (16.3) | -0.6 (10.6)
  Change at Month 48: number analyzed (Participants) | 130 | 37
  Change at Month 48 | -1.4 (16.2) | -3.8 (13.3)
  Change at Month 60: number analyzed (Participants) | 175 | 42
  Change at Month 60 | -1.7 (18.8) | -4.3 (14.1)

16. Secondary Outcome: Central Corneal Endothelial Cell Density (ECD) by Visit
Description: The endothelium maintains corneal hydration and reduced cell density can disrupt vision. Central endothelial cell counts were assessed using non-contact specular microscopy. Specular images were taken of the corneal endothelium and submitted to a reading center in order to standardize readings across all sites and optimize reading reliability. Baseline through Month 24 data were derived from COMPASS trial. A higher cell density indicates improvement. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Baseline, Month 3, 6, 12, 24, 36, 48, 60 postoperative
Population: All subject eyes for which data was available at the visit
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 214 | 67
cells/mm2
  Baseline | 2432.6 (369.7) | 2434.5 (319.6)
  Month 3: number analyzed (Participants) | 210 | 65
  Month 3 | 2199.2 (445.5) | 2227.0 (422.4)
  Month 6: number analyzed (Participants) | 211 | 64
  Month 6 | 2195.9 (431.4) | 2209.2 (412.2)
  Month 12: number analyzed (Participants) | 207 | 66
  Month 12 | 2194.3 (448.6) | 2210.9 (383.8)
  Month 24: number analyzed (Participants) | 213 | 67
  Month 24 | 2142.6 (423.3) | 2218.9 (376.0)
  Month 36: number analyzed (Participants) | 11 | 5
  Month 36 | 2148.1 (382.7) | 2258.0 (338.9)
  Month 48: number analyzed (Participants) | 116 | 33
  Month 48 | 1992.9 (460.8) | 2303.2 (334.5)
  Month 60: number analyzed (Participants) | 163 | 40
  Month 60 | 1931.2 (517.5) | 2189.1 (375.6)

17. Secondary Outcome: Number of Subjects With CyPass Device Malposition, Dislodgement or Movement
Description: Device position was a qualitative and subjective assessment by the investigator and evaluated based on visible number of rings of the device under the gonioscopic exam. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint. This outcome measure was prespecified for Cataract Surgery + CyPass arm only.
Time Frame: Up to 60 months postoperatively
Population: Total number of subjects in the treatment group
Measure: Number; unit: subjects
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 215
subjects | 6

18. Secondary Outcome: Mean Reduction From Baseline in Intraocular Pressure (IOP)
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A higher reduction from baseline (ie, a greater postitive number) indicates greater improvement. Baseline was derived from COMPASS trial. One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Baseline, Month 36, 48, 60 postoperative
Population: All subject eyes for which data was available at the visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
mmHg
  Baseline | 24.5 (2.9) | 24.8 (3.1)
  Reduction at Month 36: number analyzed (Participants) | 155 | 46
  Reduction at Month 36 | 8.9 (4.2) | 8.2 (4.6)
  Reduction at Month 48: number analyzed (Participants) | 182 | 52
  Reduction at Month 48 | 8.4 (4.5) | 7.9 (4.1)
  Reduction at Month 60: number analyzed (Participants) | 200 | 52
  Reduction at Month 60 | 8.4 (4.0) | 8.0 (4.4)

19. Secondary Outcome: Percentage of Subjects With ≥ 20% Reduction in IOP From Baseline (COMPASS Trial) Without the Use of Ocular Hypotensive Medications
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye (study eye) contributed to the analysis. Inferential testing was not planned for this endpoint.
Time Frame: Baseline, Month 36, 48, 60 postoperative
Population: All subject eyes for which data was available at the visit
Measure: Number; unit: percentage of subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
percentage of subjects
  Month 36: number analyzed (Participants) | 159 | 46
  Month 36 | 57.9 | 41.3
  Month 48: number analyzed (Participants) | 186 | 52
  Month 48 | 50.0 | 28.8
  Month 60: number analyzed (Participants) | 200 | 53
  Month 60 | 46.0 | 32.1

20. Secondary Outcome: Percentage of Subjects Not Using Ocular Hypotensive Medication With IOP ≥ 6 mmHg and ≤ 18 mmHg
Description: as for outcome 19
Time Frame: Month 36, 48, 60 postoperative
Population: All subject eyes with data available at the visit
Measure: Number; unit: percentage of subjects
Arm/Group | Cataract Surgery + CyPass | Cataract Surgery Only
Number analyzed (Participants) | 215 | 67
percentage of subjects
  Month 36: number analyzed (Participants) | 159 | 46
  Month 36 | 54.7 | 45.7
  Month 48: number analyzed (Participants) | 186 | 52
  Month 48 | 46.2 | 30.8
  Month 60: number analyzed (Participants) | 200 | 53
  Month 60 | 44.0 | 28.3

ADVERSE EVENTS:
Time Frame: Study enrollment through study completion (Month 60)
Description: This analysis population includes all enrolled subjects. Safety was assessed at each visit.
Groups:
- CyPass Micro-Stent + Cataract Surgery (Study Eye): All eyes implanted with CyPass Micro-Stent at the conclusion of cataract surgery. At risk population is reported in units of eye.
- Cataract Surgery Only (Study Eye): All eyes wherein cataract surgery occurred. At risk population is reported in units of eye
- CyPass Micro-Stent + Cataract Surgery (Systemic): All subjects implanted with CyPass Micro-Stent at the conclusion of cataract surgery (non-study eye or not eye-related).
- Cataract Surgery Only (Systemic): All subjects who underwent cataract surgery (non-study eye or not eye-related).
Arm/Group | CyPass Micro-Stent + Cataract Surgery (Study Eye) | Cataract Surgery Only (Study Eye) | CyPass Micro-Stent + Cataract Surgery (Systemic) | Cataract Surgery Only (Systemic)
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/67 | 2/215 | 1/67
Serious Adverse Events (participants affected / at risk) | 2/215 | 1/67 | 17/215 | 5/67
Other Adverse Events (participants affected / at risk) | 43/215 | 10/67 | 0/215 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CyPass Micro-Stent + Cataract Surgery (Study Eye) (N=215) | Cataract Surgery Only (Study Eye) (N=67) | CyPass Micro-Stent + Cataract Surgery (Systemic) (N=215) | Cataract Surgery Only (Systemic) (N=67)
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 2 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Conjunctival bleb (Eye disorders) | 0 | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 1
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CyPass Micro-Stent + Cataract Surgery (Study Eye) (N=215) | Cataract Surgery Only (Study Eye) (N=67) | CyPass Micro-Stent + Cataract Surgery (Systemic) (N=215) | Cataract Surgery Only (Systemic) (N=67)
Visual acuity reduced (Eye disorders) | 24 | 4 | 0 | 0
Visual field tests abnormal (Investigations) | 22 | 6 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT02700984/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02700984/SAP_001.pdf